CLINICAL TRIAL: NCT03244046
Title: Somatic Experiencing for Patients With Low Back Pain and Comorbid Posttraumatic Stress Disorder: A Randomized Controlled Trial
Brief Title: Low Back Pain and Comorbid Posttraumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern Denmark (Other)
Collaborators: Spine Centre of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tonny Elmose Andersen, phd., Associate Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT2016PTSD
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Low Back Pain; Posttraumatic Stress Disorder
Keywords: Low Back pain; Pain; Posttraumatic Stress Disorder; PTSD; Somatic Experiencing; SE
MeSH Terms: conditions — Low Back Pain; Stress Disorders, Post-Traumatic; Pain | interventions — Psychotherapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy (Phys) (Active Comparator): 12 sessions of guided physiotherapy for low back pain. Cognitive Behavioral Therapeutic elements included targeting Fear Avoidance Beliefs.
  Interventions: Behavioral: Physiotherapy
- Somatic Experiencing + phys (Experimental): 12 sessions of psychotherapy (somatic experiencing) and 12 sessions of guided physiotherapy for low back pain. Cognitive Behavioral Therapeutic elements included targeting Fear Avoidance Beliefs.
  Interventions: Behavioral: Psychotherapy; Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — The SE intervention followed the nine-step model as outlined by Peter Levine (2010) and involved gradually eliciting awareness of body sensations associated with the traumatic event. By the process of 'titration', patients were gradually encouraged to access somatic activation, feelings and body sensations as means to restore equilibrium to the autonomic nervous system and thereby alleviate hyperarousal, re-experiencing and avoidance of trauma-related experiences and thoughts.
  Other Names: Somatic Experiencing (SE)
  Arms: Somatic Experiencing + phys
Behavioral: Physiotherapy — This treatment consisted of supervised exercises for low back pain delivered in 12 sessions and performed by physiotherapists in the center according to the European guidelines for the management of chronic low back pain (Airaksinen, et al., 2006).

SUMMARY:
The aim is to test whether the psychotherapeutic intervention Somatic Experiencing targeting Post Traumatic Stress Disorder (PTSD) symptoms will have an additional positive effect on the outcomes of guided physiotherapy against chronic back pain development.

DETAILED DESCRIPTION:
Introduction: Patients with low back pain after injuries often demonstrate symptoms of PTSD measured via the Harvard Trauma Questionnaire Scale (HTQ). It has been found that PTSD and pain may maintain each other.

Methods: Thousand consecutive patients with Low Back Pain (LBP) referred to the Spine Center are screened for PTSD. It is expected that 140 patients will meet the inclusion criteria and be randomized to Guided Physiotherapy or to Guided Physiotherapy plus 12 psychotherapeutic sessions, that will include the shock-trauma method 'Somatic Experiencing'.

Effect parameters are: Pain, daily function, EuroQOL and (HTQ), anxiety and depression, fear avoidance (Tampa Scale for Kinesiophobia) and pain catastrophizing (PCS) on entry, and at 6/12 months.

ELIGIBILITY:
Inclusion Criteria:

* Back pain: from 1/2 Y duration or longer
* Trauma according to HTQ

Exclusion Criteria:

* Planned surgery, comorbid psychiatry (except PTSD and mild to moderate depression), personality disorders, drug or medical abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-01-05 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire (RMDQ; Roland & Morris, 1983) | Change from baseline to 6 months follow-up
  The RMDQ is a self-reported outcome measuring the level of disability related to low back pain. The level of disability was measured on 23 statements covering six different domains: physical ability/activity, sleep/rest, psychosocial level of functioning, household management, eating, and pain frequency. Each statement was scored 1 if the patient felt that the statement was descriptive of their circumstances and scored 0 if not. The total RMDQ score ranges from 0 (no disability) to 23 (maximal disability). Scores were converted to percentages with 24 corresponding to 100% disability.
Harvard Trauma Questionnaire part IV (Mollica, Caspi-Yavin, Bollini, & Truong, 1992) | Change from baseline to 6 months follow-up
  The Harvard Trauma Questionnaire consists of 17 items with a 4-point Likert scale (1 = not at all to 4 = very often). The 17 items relate to PTSD's core clusters within the Diagnostic and Statistical Manual of Mental Disorders (APA, 1994), 4th Edition (DSM-IV): avoidance (7 items), re-experiencing (5 items), and hyperarousal (5 items). An item was deemed to be positively endorsed if scores were ≥ 3. The Harvard Trauma Questionnaire follows the diagnostic criteria for the PTSD diagnosis according to the DSM-IV. The scale thus makes it possible to measure both the severity of symptoms and to estimate the prevalence of possible PTSD. Following the DSM-IV, a possible PTSD diagnosis was proposed if participants reported at least one re-experiencing symptom, three avoidance symptoms, and two hyperarousal symptoms.

SECONDARY OUTCOMES:
Pain intensity | baseline, 3, 6 and 12 months
  Pain intensity was measured as the average score of three 11-point Likert scales measuring peak pain intensity, average pain intensity over the past 2 weeks as well as current pain intensity (Manniche, Asmussen, Lauritsen, Vinterberg, et Kreiner, 1994). Each scale measured pain intensity on a 0-10 numerical rating scale (NRS: Jensen, Karoly, & Braver, 1986) with 0 defined as no pain and 10 as the worst imaginable pain.
The Pain Catastrophizing Scale (Sullivan, Bishop, & Pivik, 1995) | baseline, 3, 6 and 12 months
  The Pain Catastrophizing Scale (Sullivan, Bishop, & Pivik, 1995) was used to measure catastrophic thinking related to pain. Its instructions ask participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on a 5-point Likert scale with (0 = not at all, 4 = all the time). A scale sum score was calculated from all items, with a high score indicating a high level of pain catastrophizing.
the Tampa Scale for Kinesiophobia (TSK: Kori, Miller, & Todd, 1990). | baseline, 3, 6 and 12 months
  Fear of re-injury due to movement was measured with the Tampa Scale for Kinesiophobia (TSK: Kori, Miller, & Todd, 1990). TSK is a 17-item scale assessing fear of movement on a 4-point Likert scale ranging from 17 to 68 with higher scores indicating higher levels of kinesiophobia. The scale is commonly used in diverse chronic pain samples and has good construct and predictive validity (Vlaeyen, Kole-Snijders, Boeren, & van Eek, 1995).
Anxiety and Depression (Hospital and Anxiety Depression Scale, HADS) | baseline, 3, 6 and 12 months
  The scale consists of 14 items, seven relating to anxiety (HADS-A) and seven to depression (HADSD) with responses ranging from 0 (no symptoms) to 3 (maximum impairment). In the present study, we used a subscale cut-off of 8 in order to include all possible cases of anxiety or depression, as suggested by Zigmond and Snaith (1983).

CONTACTS AND LOCATIONS:
Overall Officials: Berit Schiøttz-Christensen, professor, Study Director — Spine Center South

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen TE, Ellegaard H, Schiottz-Christensen B, Manniche C. Somatic experiencing(R) for patients with low back pain and comorbid posttraumatic stress disorder - protocol of a randomized controlled trial. BMC Complement Altern Med. 2018 Nov 22;18(1):308. doi: 10.1186/s12906-018-2370-y. PMID 30466429